CLINICAL TRIAL: NCT06527144
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase II Clinical Trial of the Efficacy and Safety of Inhaled TQC3721 Suspension in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Clinical Trial of TQC3721 Suspension for Inhalation in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC3721-II-03
Record Dates: First submitted 2024-07-24; First posted 2024-07-30 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3mg TQC3721 Suspension for Inhalation (Twice a day) (Experimental): Two syringes of TQC3721 suspension for inhalation (1ml:1.5mg), twice a day for 4 weeks.
  Interventions: Drug: 3mg TQC3721 Suspension for Inhalation
- 6mg TQC3721 Suspension for Inhalation (Twice a day) (Experimental): one syringe of TQC3721 suspension for inhalation（1ml:6mg）and one TQC3721 suspension placebo for inhalation (1ml:0mg), twice a day for 4 weeks.
  Interventions: Drug: 6mg TQC3721 Suspension for Inhalation
- Placebo for TQC3721 Suspension for Inhalation (Twice a day) (Placebo Comparator): Two syringes of placebo for TQC3721 suspension for inhalation (1ml:0mg), twice a day for 4 weeks.
  Interventions: Drug: Placebo TQC3721 suspension for inhalation

INTERVENTIONS:
Drug: 3mg TQC3721 Suspension for Inhalation — TQC3721 suspension for inhalation is target inhibitor.
  Arms: 3mg TQC3721 Suspension for Inhalation (Twice a day)
Drug: 6mg TQC3721 Suspension for Inhalation — TQC3721 suspension for inhalation is target inhibitor.
  Arms: 6mg TQC3721 Suspension for Inhalation (Twice a day)
Drug: Placebo TQC3721 suspension for inhalation — Placebo without active drug substance.
  Arms: Placebo for TQC3721 Suspension for Inhalation (Twice a day)

SUMMARY:
To evaluate the efficacy and safety of TQC3721 Suspension for Inhalation in patients with moderate to severe Chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent before the test and fully understand the test content, process and possible adverse reactions.
* Male and female subjects aged 40 to 80 years old (including the cut-off value).
* Body mass index (BMI) in the range of 18-30kg/m2 (including the critical value)
* Subjects have no pregnancy plan and voluntarily use effective contraception for at least 1 month from screening to the last use of the study drug.
* Diagnosed as a COPD patient according to the The Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2024 criteria.
* Able to conduct acceptable and reproducible lung function tests.
* COPD clinical stability within the 4 weeks prior to screening visit (V1 visit) and between V1 visit and V2 visit.
* Smoking history ≥ 10 pack years.

Exclusion Criteria:

* History of life-threatening COPD, including admission to the intensive care unit and/or the need for intubation.
* Screening for COPD acute exacerbations that require systemic hormone therapy prior to the visit.
* Screening for hospitalization history due to COPD within the first 6 months.
* Use antibiotics for respiratory tract infections within 6 weeks prior to screening or randomization visit.
* Chest computed tomography (CT) revealed clinically significant abnormalities and concluded that the abnormalities were not caused by COPD.
* Previous lung resection or lung reduction surgery.
* Pulmonary rehabilitation treatment.
* Previously received TQC3721 treatment.
* Patients who received immunotherapy within the first 4 weeks of the screening period.
* The patient has a history of diseases that are currently beyond their control.
* History or current evidence of cardiovascular disease with clinical significance.
* History of cured or untreated malignant tumors in any organ or system within the past 5 years.
* Screening for clinically significant safety laboratory test outliers determined by the researcher during the visit.
* Those who require oxygen therapy or intermittent oxygen therapy.
* Receive attenuated live vaccine within 28 days prior to randomization, inactivated vaccine within 7 days, or study.
* Planned vaccine recipients during the period.
* Individuals who have participated in any drug or medical device clinical trials prior to screening.
* Researchers believe that there are other situations that are not suitable for participation in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-03-06 (Actual)

PRIMARY OUTCOMES:
Change of the maximum value of Forced Expiratory Volume in the first second (FEV1) | From baseline to four weeks after treatment
  Change of the maximum value of FEV1 was determined from baseline to four weeks after treatment.

SECONDARY OUTCOMES:
Change of the mean value of FEV1 | From baseline to four weeks after treatment
  Compared with baseline, the mean value of FEV1 was changed within 3 hours and 12 hours after morning medication at 4 weeks of treatment.
Changes in peak FEV1 values,trough FEV1 values, mean value within 3 hours after administration | From baseline to two weeks after treatment
  Compared with baseline, Changes in peak FEV1 values,trough FEV1 values, mean value within 3 hours after administration after 2 weeks of treatment.
Rescue medication | From baseline to four weeks after administration
  Frequency of Rescue medication use during the study compared to placebo group
Adverse Events (AE) | From baseline to safety visit (about 5 weeks after first dosing).
  The number, frequency, incidence, and severity of adverse events, serious adverse events, and adverse events associated with investigational drugs (including investigational drugs and control drugs), as well as abnormal laboratory indicators were evaluated.
Changes in the peak value of FEV1，mean value of FEV1 within 3 hours and 12 hours after administration | From baseline to 1day after treatment
  Compared with baseline, changes in the peak value of FEV1 after 1 day of treatment, and the mean value of FEV1 within 3 hours and 12 hours after administration.
Changes of FEV1 at each time point | From baseline to 1day after treatment
  Changes in series FEV1 at each time point within 12 hours after morning administration on day 1 of treatment (after first dosing) compared to baseline.
Changes in peak value of FEV1 and the mean value of FEV1 within 3 hours and 12 hours | From 1day after treatment to 4 weeks after treatment
  To evaluate the change in FEV1 peak value and FEV1 mean value within 3 hours and 12 hours after 4 weeks of treatment compared with 1 day of treatment (after first administration)
Changes in Morning Valley FEV1 | From baseline to four weeks after treatment
  Changes in Morning Valley FEV1 after 4 weeks of treatment compared with baseline
Changes in Modified Medical Research Council (mMRC) Dyspnea Scale Score | Changes in mMRC score after 2 and 4 weeks of treatment compared with baseline
  mMRC Dyspnea Scale Score's total score is 0-4 points, with the higher score meaning the more severe symptoms.
Chronic obstructive pulmonary disease Assessment Test (CAT) | Changes in CAT assessment after 2 and 4 weeks of treatment compared with baseline
  There are 8 questions in the CAT, and each question is scored 0-5 points, with the higher score meaning the more severe symptoms
St. George's Respiratory Questionnaire (SGRQ) | Changes in SGRQ after 2 and 4 weeks of treatment compared with baseline
  SGRQ has three parts: symptoms, abilities, and effects, and is used to comprehensively measure the physical, mental, and social status of COPD patients.
Basic Dyspnea Index (BDI) | Changes in BDI after 2 and 4 weeks of treatment compared with baseline.
  BDI has three levels: functional impairment, magnitude of task, and magnitude of effort. Each level is rated from 0 (severe) to 4(No damage).
Transitional Dyspnea Index (TDI) | Changes in TDI after 2 and 4 weeks of treatment compared with baseline
  TDI has three levels:changes in functional impairment, changes in magnitude of task, changes in magnitude of effort,. Scores in each area range from -3 (significant deterioration) to 0 (no change) to +3 (significant improvement).

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - Fu Yang People'S Hospital, Fuyang, Anhui
  - ChongQing University Fuling Hospital, Chongqing, Chongqing Municipality
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Zunyi Medical University Affiliated Hospital, Zunyi, Guizhou
  - Cangzhou Hospital of Integrated Tcm-Wm·Hebei, Cangzhou, Hebei
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Shangqiu First People's Hospita, Shangqiu, Henan
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - Wuxi Fifth People's Hospital, Wuxi, Jiangsu
  - Yixing People'S Hospital, Wuxi, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Siping Central People's Hospital, Siping, Jilin
  - Genertec Liaoyou Gem Flower Hospital, Panjin, Liaoning
  - Heze Municipal Hospital, Heze, Shandong
  - Shanghai JiaoTong University of medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Suining Central Hospital, Suining, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - TianJin 4th Center Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Shihezi University, Shihezi, Xinjiang
  - Wenzhou University Affiliated Second Hospital, Wenzhou, Zhejiang